CLINICAL TRIAL: NCT01001065
Title: Association of the Intrarenal Resistance Index (RI) of Transplanted Kidneys With Generalized Atherosclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Christoph Thalhammer, MD, USZ
Other Study IDs: CT-03-2009-USZ
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Renal Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Vascular ultrasound — RI ist predictive for arteriosclerosis

SUMMARY:
Cross sectional observational ultrasound study of transplanted kidneys and the carotid artery in consecutive recruited outpatients.

ELIGIBILITY:
Inclusion criteria:

* Patients after renal transplantation with stable renal function

Exclusion criteria:

* Known impairment of renal function (e.g. acute rejection)
* Known renal artery or carotid artery stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after renal transplantation with stable renal function
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2009-10; Study Completion 2010-10

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland